CLINICAL TRIAL: NCT07211165
Title: Study on the Mass Balance of [14C] Clifutinib in Chinese Male Healthy Subjects
Brief Title: Clinical Study on the Mass Balance of Clifutinib
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sunshine Lake Pharma Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HEC73543-AML-104
Record Dates: First submitted 2025-09-22; First posted 2025-10-07 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2025-09

CONDITIONS: Healthy Adult Male
Keywords: Clifutinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- [14C]Clifutinib (Experimental): On Day 1, subjects will receive a single oral dose of 40 mg/100 µCi [14C]Clifutinib
  Interventions: Drug: [14C]Clifutinib

INTERVENTIONS:
Drug: [14C]Clifutinib — The subjects are required to take the test drug on an empty stomach for at least 10 hours and without drinking water for 1 hour. After taking the drug, they should fast for 4 hours and refrain from drinking water for 1 hour.

SUMMARY:
To investigate the plasma total radioactivity PK characteristics of male healthy subjects after a single oral administration of [14C]Clifutinib, the distribution of total radioactivity in whole blood and plasma, and to determine the main excretion and metabolic pathways.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male, age: 18 - 45 years (inclusive of boundary values).
2. Weight of no less than 50 kg, and body mass index (BMI) within the range of 19 kg/m2 - 26 kg/m2 (including critical values).
3. Signed the informed consent form before the trial and fully understood the trial content, process and possible adverse reactions.
4. The subjects can communicate well with the researchers and complete the trial in accordance with the protocol.

Exclusion Criteria:

1. Those with abnormal and clinically significant findings in comprehensive physical examination, routine laboratory tests (blood routine, blood biochemistry, C-reactive protein, coagulation function, urine routine), stool routine + occult blood, thyroid function, 12-lead electrocardiogram, chest CT, abdominal B-ultrasound (liver, gallbladder, pancreas, spleen, kidney), etc.
2. Those who fail the vital sign examination and still fail after re-examination.
3. Those with abnormal and clinically significant findings in ophthalmological examination (slit lamp, intraocular pressure, fundus photography).
4. Those with abnormal and clinically significant findings in hepatitis B surface antigen, hepatitis B e antigen, anti-HCV IgG, HIV-Ag/Ab, and syphilis antibody tests, as determined by the investigator.
5. Those who have used CYP3A4 inhibitors or inducers within 30 days before the screening period, as detailed in Appendix 1.
6. Those who have used any prescription drugs, over-the-counter drugs, herbal health products, or food supplements (such as vitamins, calcium supplements) within 14 days before the screening period.
7. Those with a history of or current diseases in the musculoskeletal system, nervous and mental system, endocrine system, circulatory system, respiratory system, digestive system, urinary system, reproductive system, etc., and the investigator deems it clinically significant.
8. Those with any diseases that increase the risk of elevated blood sugar, such as a history of primary diabetes, steroid-induced diabetes, other secondary diabetes, acute or chronic pancreatitis, and the investigator deems it clinically significant.
9. Those with a history of organic heart disease, heart failure, myocardial infarction, angina pectoris, unexplained arrhythmia, torsades de pointes, ventricular tachycardia, atrioventricular block, and the investigator deems it clinically significant; those with QTcF > 450ms during the screening period.
10. Those with interstitial lung disease, severely impaired lung function, severe pulmonary fibrosis, radiation pneumonitis, drug-induced lung disease, and evidence of active pulmonary inflammation on chest CT during the screening period, and the investigator deems it clinically significant.
11. Those who have undergone major surgery within 6 months before the screening period or whose surgical incisions have not fully healed; major surgeries include but are not limited to any surgeries with significant bleeding risk, prolonged general anesthesia, or incisional biopsy or obvious traumatic injury, or surgeries that affect drug absorption, distribution, metabolism, and excretion, or those planning to undergo surgery during the study period.
12. Those with drug, environmental, food allergies or allergic constitution, or those the investigator deems may be allergic to the study drug or its excipients.
13. Those with hemorrhoids or perianal diseases with regular/ongoing bleeding, irritable bowel syndrome, inflammatory bowel disease.
14. Those with multiple factors affecting oral and drug absorption (such as inability to swallow, post-gastrointestinal resection, ulcerative colitis, symptomatic/inflammatory bowel disease, and intestinal obstruction, etc.).
15. Those with habitual constipation or diarrhea.
16. Those with lactose intolerance (those who have experienced diarrhea after drinking milk).
17. Those who are heavy drinkers or have frequently consumed alcohol within 6 months before the screening period (more than 14 units of alcohol per week, 1 unit = 360 mL of beer or 45 mL of 40% alcohol or 150 mL of wine), or those who cannot abstain from alcohol during the trial, or those with a breath alcohol test result > 0 mg/100 mL during the screening period.
18. Those who smoke more than 5 cigarettes per day or habitually use nicotine-containing products within 3 months before the screening period and cannot quit during the trial.
19. Those who have abused drugs or used soft drugs (such as marijuana) within 3 months before the screening period or hard drugs (such as cocaine, amphetamines, phencyclidine, etc.) within 1 year before the screening period, or those with positive urine drug tests during the screening period.
20. Habitual consumption of grapefruit juice or excessive tea, coffee and/or caffeine-containing beverages, and those who are unable to abstain during the trial period.
21. Workers exposed to radiation for long periods of time, or those who have had significant radiation exposure (≥2 chest/abdominal CTs or ≥3 other types of X-ray examinations) within one year prior to signing the ICF, or those who have participated in radiolabeled drug trials within one year prior to signing the ICF.
22. Those with a history of fainting at the sight of needles or blood, or those who have difficulty with blood collection or cannot tolerate venipuncture.
23. Those who have participated in other clinical trials and used other investigational drugs or devices within three months before screening or during the screening period, or those who plan to participate in other clinical trials during this study, or those who are not the subjects themselves.
24. Those who have received vaccinations within one month before screening or plan to receive vaccinations during the trial period.
25. Those who have plans to conceive or donate sperm within one year from signing the ICF to one year after receiving the investigational drug, or those who do not agree that both the subject and their spouse should take strict contraceptive measures during this period (see Appendix 3 for details).
26. Those who have lost or donated blood of 400 mL or more within three months before the screening period, or those who have received blood transfusions within one month.
27. Those who are considered unsuitable for participation in the trial by the investigator for other reasons, or those who withdraw from the trial for their own reasons.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2025-09-29 (Actual); Primary Completion 2025-11-05 (Actual); Study Completion 2025-11-12 (Actual)

PRIMARY OUTCOMES:
AUC0-∞ | From Day 1 of dosing to the Day 85 after dosing
  Investigate the plasma total radioactivity PK characteristics of male healthy subjects after a single oral administration of [14C] Clifutinib
Tmax | From Day 1 of dosing to the Day 85 after dosing
  Investigate the plasma total radioactivity PK characteristics of male healthy subjects after a single oral administration of [14C] Clifutinib
Cmax | From Day 1 of dosing to the Day 85 after dosing
  Investigate the plasma total radioactivity PK characteristics of male healthy subjects after a single oral administration of [14C] Clifutinib
Percentage of metabolites in plasma relative to total exposure AUC (% AUC) | From Day 1 of dosing to the Day 85 after dosing
  Investigate the distribution of total radioactivity in plasma of male healthy subjects after a single oral administration of [14C] Clifutinib.
The total radioactivity | From Day 1 of dosing to the Day 85 after dosing
  Quantitative analysis was conducted on the total radioactivity in the feces and urine of male health subjects after oral administration of [14C] Clifutinib, to obtain the data on human recovery rate and determine the main excretion pathway.
Identification of major metabolites in plasma, urine, and fecal samples | From Day 1 of dosing to the Day 85 after dosing
  Obtain the radioactive metabolite profiles in plasma, urine and feces of male healthy subjects after oral administration of [14C]Clifutinib, identify the main metabolites, and determine the metabolic and elimination pathways.

SECONDARY OUTCOMES:
AUC0-∞ | From Day 1 of dosing to the Day 85 after dosing
  The validated liquid chromatography-tandem mass spectrometry (LC-MS/MS) method was used to quantitatively analyze the concentrations of Clifutinib, its metabolite (M3), and other metabolites (if applicable) in plasma, thereby obtaining the corresponding pharmacokinetic parameters.
Tmax | From Day 1 of dosing to the Day 85 after dosing
  The validated liquid chromatography-tandem mass spectrometry (LC-MS/MS) method was used to quantitatively analyze the concentrations of Clifutinib, its metabolite (M3), and other metabolites (if applicable) in plasma, thereby obtaining the corresponding pharmacokinetic parameters.
Cmax | From Day 1 of dosing to the Day 85 after dosing
  The validated liquid chromatography-tandem mass spectrometry (LC-MS/MS) method was used to quantitatively analyze the concentrations of Clifutinib, its metabolite (M3), and other metabolites (if applicable) in plasma, thereby obtaining the corresponding pharmacokinetic parameters.
Frequency, type and severity of adverse events/serious adverse events; changes in vital signs, 12-lead ECGs, laboratory tests, etc. | From Day 1 of dosing to the Day 85 after dosing
  Observation of the safety profile in male healthy subjects after a single administration of [14C] Clifutinib

CONTACTS AND LOCATIONS:
Locations (1):
- Affiliated hospital of Jiangnan University, Wuxi, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No